CLINICAL TRIAL: NCT05663216
Title: Determinants of Vascular Leakage During Systemic Inflammatory Response Syndrome
Acronym: SIRS-PERM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220418
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Systemic inflammatory response syndrome; Vascular leakage; Capillary leakage; fluid balance
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Six ml of blood will be sampled at Day 0 (beginning of the SIRS), D1, D3, D7
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling — 6 ml blood sampling at Day 0, 1, 3, 7. Broncho-alveolar sampling, if performed in routine care.

SUMMARY:
BACKGROUND Controlling vascular leakage, which is independently associated with mortality during Sepsis and cardiogenic shock, may be a promising approach during systemic inflammatory response syndrome (SIRS). During a collaborative work between La Pitié-Salpêtrière intensive care unit (ICU) and the unit INSERM U1050 (National Institute oh Health and medical Research), we identified 38 genes associated with capillary leakage during systemic inflammation response syndrome (SIRS) in humans. The aim of this study is to evaluate their possible implication in vascular hyperpermeability associated with

METHODS SIRS-PERM is a prospective multicenter cohort study, testing the correlation between the plasma and broncho-alveolar levels of proteins isolated from our first screening, and the level of vascular leakage during SIRS. All patients admitted in the European Georges-Pompidou or La Pitié-Salpêtrière ICU and presenting a SIRS will be eligible for inclusion. Plasma samples will be collected at day 0, D1, D3 and D7, as well as broncho-alveolar lavage samples if clinically indicated. Concentration of each protein will be determined by ELISA in those samples. A statistical association will be then tested between each protein concentration and, for each time-point, the level of capillary leakage (daily weight and fluid balance, extra-vascular lung water index and pulmonary permeability index measured by transpulmonary thermodilution), and ARDS (acute respiratory distress syndrome) severity (PaO2/FiO2 ratio, Murray score and pulmonary compliance). Its link with hemodynamic status, the level of multiple organ failure, and vital status at day 30, will be also assessed. Basing the calculation of the sample size on the variations of VEGF (Vascular endothelial growth factor) expression in our first screening cohort, we calculated a sample size of 180 patients for this study, for a total duration of the study of 5 years.

IMPLICATIONS: SIRS-PERM will assess the determinants of capillary leakage during SIRS. It may thus provide a better understanding of the pathophysiology of this disease, with the goal to isolate new markers of severity, as well as new therapeutic targets to treat it. Modulating specifically capillary leakage is indeed a totally new approach during this pathology.

DETAILED DESCRIPTION:
1. Intervention Six ml of blood will be sampled at Day 0 (beginning of the SIRS), D1, D3, D7. Concentrations of candidate proteins will be determined in the plasma by ELISA, and the link between each concentration and each outcome analyzed.

   Additionally, broncho-alveolar lavage will be analyzed in the same way, if performed for the routine care of the patient.
2. Statistical analysis

The link between plasma and alveolar levels of each protein and each outcome will be evaluated, using Mann-Whitney U-test and one-way ANOVA for categorical variables (for example comparison of protein X plasma level between survivors or nonsurvivors at 30 days), and Pearson's correlation for continuous variables (for example link between protein X plasma level and daily fluid balance at each time point).

Sample size calculation. Plasma and pulmonary concentrations of each protein that we will study have never been described during SIRS. Based on our first screening cohort patients with severe capillary leakage had a difference in VEGF plasma concentration of 15.5 pg/ml, with a standard deviation of 32 pg/ml. Basing the calculation on this parameter, with an alpha risk of 5% and a power of 90%, a sample size of 180 patients would provide 90% chances to find a statistical link between one protein concentration and the outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the European Georges Pompidou Hospital or La Pitié-Salpêtrière ICU, and exhibiting a systemic inflammatory response syndrome (SIRS), characterized by the following items:

  * Temperature > 38°C ou <36°C
  * Heart rate >90/min
  * Respiratory rate >20/min or PaCO2<32mmHg
  * White cell count > 12 000/mm3 ou < 4 000/mm3

Exclusion Criteria:

* Age <18 years
* Decline to participate
* Pregnancy
* Cirrhosis Child-Pugh > B
* Denutrition with BMI<15kg/m2
* Nephrotic syndrome
* Persons deprived of their liberty by a judicial or administrative decision (guardianship or tutelage measure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in the European Georges Pompidou Hospital or La Pitié-Salpêtrière ICU, and exhibiting a systemic inflammatory response syndrome (SIRS)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Fluid balance from Day 0 to day 3 (ml/kg of initial body weight). | Between Day 0 and Day 3
  The fluid balance, routinely monitored in ICU, represents fluid intakes (perfusion, oral intakes,..) - fluid losses (diuresis, diarrhea,...)

SECONDARY OUTCOMES:
Fluid balance (ml/kg of initial body weight). | Day 1, Day 3, Day 7
  The fluid balance, routinely monitored in ICU, represents fluid intakes (perfusion, oral intakes,..) - fluid losses (diuresis, diarrhea,...)
Extra-vascular lung water index | Day 0, Day 1, Day 3, Day 7
  Extra-vascular lung water index (EVLWi, ml/kg) and pulmonary vascular permeability index measured by transpulmonary thermodilution at corresponding time-points
SOFA score | Day 0, Day 1, Day 3, Day 7,
  Association between circulating candidate proteins, the immune-inflammatory profile of the patients and SOFA score (Sepsis-related Organ Failure Assessment), score values between 0-24, higher scores mean a worse outcome
Serum albuminemia | Day 0, Day 1, Day 3, Day 7,
  Serum albuminemia in g/L
Catecholamine-free days | Day 0, Day 1, Day 3, Day 7, Day 30
  Number of days alive without receiving any catecholamine
Ventilatory-free days | Day 0, Day 1, Day 3, Day 7, Day 30
  Number of days alive without receiving any mechanical ventilation, invasive or non-invasive
Renal replacement therapy-free Number of days alive without receiving any renal replacement therapy | Day 0, Day 1, Day 3, Day 7, Day 30
  Number of days alive without receiving any renal replacement therapy
Mortality | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Brechot, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Adult Medical-Surgical Intensive Care Unit, Necker Hospital of the Sick Children, Paris
  - Medical Intensive Care Unit, Georges Pompidou European Hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
All deidentified individual participant data collected for our study "SIRS-PERM" will be shared beginning with publication with no end date. These data will be available to researchers to who provide a methodologically sound proposal for the purposes of achieving specific aims outlined in that proposal. Proposals should be directed to the corresponding author via email: nicolas.brechot@aphp.fr and will be reviewed by the senior authors of the study. Requests to access data to undertake hypothesis-driven research will not be unreasonably withheld. To gain access, data requesters will need to sign a data access agreement and to confirm that data will only be used for the agreed purpose for which access was granted.